CLINICAL TRIAL: NCT05928650
Title: Comparison of Menstrual Function Among Sprinters, Long Marathon Runners, and Non-athletic Females: An Observational Study
Brief Title: Comparison of Menstrual Function Among Sprinters, Long Marathon Runners, and Non-Athletic Females
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Doaa A. Osman, Assistant Professor, Cairo University
Other Study IDs: P.T.REC/012/004550
Record Dates: First submitted 2023-06-26; First posted 2023-07-03 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Menstruation Disturbances
Keywords: Menstrual function; Serum estradiol levels; Sprinters; Long Marathon Runners; Non-Athletic Females
MeSH Terms: conditions — Menstruation Disturbances

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Sprinters: Sprinters
  Interventions: Other: Evaluation of menstrual function
- Long marathon runners: Long marathon runners
  Interventions: Other: Evaluation of menstrual function
- Non-athletic Females: Non-athletic Females
  Interventions: Other: Evaluation of menstrual function

INTERVENTIONS:
Other: Evaluation of menstrual function — Evaluation of serum estradiol levels and menstrual history characteristics between sprinters, long marathon runners and non-athletes.

SUMMARY:
The purpose of this study is to compare between sprinters and long marathon in menstrual characteristics and serum estradiol level.

DETAILED DESCRIPTION:
Menstrual function and dysfunction conversations have long been stigmatized both in the general population and in sport settings (O'Flynn, 2006). However, Discussions of menstruation in the sport context often focuses on the impact of physical menstrual symptoms and dysfunction on activities such as training and sport performance (Bruinvels et al., 2016; Knowles et al., 2019). In addition, no study had been compare between sprinters and long-marathon runners in menstrual characteristics and estradiol level. Therefore, the purpose of this study to compare between sprinters and long marathon in menstrual characteristics and serum estradiol level.

ELIGIBILITY:
Inclusion Criteria:

* Virginal females.
* Their age ranged from 16 to 19years.
* All females had the same socio-economic status.

For athletic groups only:

* They have been starting the practice of sport at least one year before the onset of menarche.

Exclusion Criteria:

* Females who had been used oral contraceptives or any hormonal treatment in the previous six months.
* Smoking.
* History of chronic disease.
* Having any psychiatric problems.

For athletic groups only:

* injured females who were absent from training for at least three months.

Ages: 16 Years to 19 Years | Sex: Female
Age Groups: Child, Adult
Gender Based: Yes — Participant eligibility is based on self-representation of gender identity.
Study Population: Egyptian sprinters, long marathon runners, and non-athletic females
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
serum estradiol level | 3 months
  Blood samples were obtained on the 2nd day of the menstrual cycle at 10.00 a.m. following overnight fasting and rest. The athletic females were instructed to refrain from performing strenuous exercise on the day of sampling. Blood samples were separated and stored at -80°C till analysis of serum estradiol levels. Serum estradiol levels were measured to evaluate the menstrual function. The manufacturer indicated the following reference intervals for healthy females: Estradiol 40-350 pg/ml.
Menstrual history characteristics | 3 months
  The age at menarche (in years), the number of menstrual cycles in the past year, and the length of menstrual cycles (in days) were collected through a self-administered questionnaire to evaluate the menstrual status of each female participant.
Age of participation to sport | 3 months
  It was taken in years from each female athlete through a self-administered questionnaire.
Weekly training workload | 3 months
  It was taken in hours per week from each female athlete through a self-administered questionnaire.
Training experience | 3 months
  The training experience of the athlete was then calculated by subtracting her age of participation in sport from her chronological age.

CONTACTS AND LOCATIONS:
Overall Officials: Doaa Osman, Principal Investigator — Department of Physical Therapy for Woman's Health, Faculty of physical therapy, Cairo University, Giza, Egypt.
Locations (1):
- Faculty of Physical therapy, Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No